CLINICAL TRIAL: NCT00365716
Title: A Placebo-Controlled, Dose-Ranging Study of Quadrivalent HPV Virus-Like Particle (VLP) Vaccine in 16- to 23-Year-Old Women
Brief Title: Dose-Ranging Study of Quadrivalent Human Papillomavirus (HPV) (Types 6,11,16,18) L1 Virus-Like Particle (VLP) Vaccine (V501-007)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-007; 2006_516
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Papillomavirus Infections; Genital Diseases, Female
Keywords: HPV 6/11/16/18 infection and related genital disease
MeSH Terms: conditions — Papillomavirus Infections; Genital Diseases, Female | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine (Experimental): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 1 received a 20/40/40/20 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  Interventions: Biological: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 (Experimental): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 2 received a 40/40/40/40 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  Interventions: Biological: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 (Experimental): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 3 received a 80/80/40/80 formulation of quadrivalent human papillomavirus (qHPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  Interventions: Biological: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80
- Placebo (mcg) (Aluminum Adjuvant) 225 (Experimental): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 4 received placebo containing 225 mcg of aluminum adjuvant per dose at Day 1, Month 2, and Month 6.
  Interventions: Biological: Placebo (mcg) (Aluminum Adjuvant)225
- Placebo (mcg) (Aluminum Adjuvant) 450 (Experimental): The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 5 received placebo containing 450 mcg of aluminum adjuvant per dose at Day 1, Month 2, and Month 6.
  Interventions: Biological: Placebo (mcg) (Aluminum Adjuvant) 450

INTERVENTIONS:
Biological: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 — 20/40/40/20 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  Other Names: V501
  Arms: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine
Biological: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 — 40/40/40/40 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  Other Names: V501
  Arms: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40
Biological: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 — 80/80/40/80 formulation of quadrivalent human papillomavirus (qHPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  Other Names: V501
  Arms: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80
Biological: Placebo (mcg) (Aluminum Adjuvant)225 — placebo containing 225 mcg of aluminum adjuvant per dose at Day 1, Month 2, and Month 6.
  Arms: Placebo (mcg) (Aluminum Adjuvant) 225
Biological: Placebo (mcg) (Aluminum Adjuvant) 450 — placebo containing 450 mcg of aluminum adjuvant per dose at Day 1, Month 2, and Month 6.
  Arms: Placebo (mcg) (Aluminum Adjuvant) 450

SUMMARY:
This study was conducted in 2 parts. Part A was a randomized, double-blind, placebo-controlled, multicenter, sequential dose-escalating evaluation. Part B was a randomized, double-blind (operating under in-house blinding procedures), placebo-controlled, multicenter, dose-ranging study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females 16 to 23 years of age
* Not pregnant at enrollment and must have agreed to use effective contraception through Month 7 of the study
* Lifetime history of 0 to 4 male sexual partners (individuals with whom penetrative sexual intercourse occurred)

Exclusion Criteria:

* No prior receipt of an Human Papillomavirus (HPV) vaccine
* No receipt of inactivated or recombinant vaccines within 14 days prior to enrollment or receipt of live vaccines within 21 days prior to enrollment
* No prior abnormal Pap test showing squamous intraepithelial lesion (SIL) or biopsy showing cervical intraepithelial neoplasia (CIN)
* No prior history of genital warts or treatment for genital warts

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1158 (Actual)
Dates: Start 2000-05; Primary Completion 2004-05 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Ault KA, Giuliano AR, Wheeler CM, Koutsky LA, Malm C, Lehtinen M, Skjeldestad FE, Olsson SE, Steinwall M, Brown DR, Kurman RJ, Ronnett BM, Stoler MH, Ferenczy A, Harper DM, Tamms GM, Yu J, Lupinacci L, Railkar R, Taddeo FJ, Jansen KU, Esser MT, Sings HL, Saah AJ, Barr E. Prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in young women: a randomised double-blind placebo-controlled multicentre phase II efficacy trial. Lancet Oncol. 2005 May;6(5):271-8. doi: 10.1016/S1470-2045(05)70101-7. PMID 15863374
- [Background] Villa LL, Ault KA, Giuliano AR, Costa RL, Petta CA, Andrade RP, Brown DR, Ferenczy A, Harper DM, Koutsky LA, Kurman RJ, Lehtinen M, Malm C, Olsson SE, Ronnett BM, Skjeldestad FE, Steinwall M, Stoler MH, Wheeler CM, Taddeo FJ, Yu J, Lupinacci L, Railkar R, Marchese R, Esser MT, Bryan J, Jansen KU, Sings HL, Tamms GM, Saah AJ, Barr E. Immunologic responses following administration of a vaccine targeting human papillomavirus Types 6, 11, 16, and 18. Vaccine. 2006 Jul 7;24(27-28):5571-83. doi: 10.1016/j.vaccine.2006.04.068. Epub 2006 May 15. PMID 16753240
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Paavonen J, Iversen OE, Olsson SE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, Krogh Gv, Lehtinen M, Malm C, Tamms GM, Giacoletti K, Lupinacci L, Railkar R, Taddeo FJ, Bryan J, Esser MT, Sings HL, Saah AJ, Barr E. High sustained efficacy of a prophylactic quadrivalent human papillomavirus types 6/11/16/18 L1 virus-like particle vaccine through 5 years of follow-up. Br J Cancer. 2006 Dec 4;95(11):1459-66. doi: 10.1038/sj.bjc.6603469. Epub 2006 Nov 21. PMID 17117182
- [Background] Barr E, Gause CK, Bautista OM, Railkar RA, Lupinacci LC, Insinga RP, Sings HL, Haupt RM. Impact of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle vaccine in a sexually active population of North American women. Am J Obstet Gynecol. 2008 Mar;198(3):261.e1-11. doi: 10.1016/j.ajog.2007.09.001. PMID 18313445
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] Perez G, Lazcano-Ponce E, Hernandez-Avila M, Garcia PJ, Munoz N, Villa LL, Bryan J, Taddeo FJ, Lu S, Esser MT, Vuocolo S, Sattler C, Barr E. Safety, immunogenicity, and efficacy of quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like-particle vaccine in Latin American women. Int J Cancer. 2008 Mar 15;122(6):1311-8. doi: 10.1002/ijc.23260. PMID 18000825
- [Background] Olsson SE, Villa LL, Costa RL, Petta CA, Andrade RP, Malm C, Iversen OE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, von Krogh G, Lehtinen M, Paavonen J, Tamms GM, Giacoletti K, Lupinacci L, Esser MT, Vuocolo SC, Saah AJ, Barr E. Induction of immune memory following administration of a prophylactic quadrivalent human papillomavirus (HPV) types 6/11/16/18 L1 virus-like particle (VLP) vaccine. Vaccine. 2007 Jun 21;25(26):4931-9. doi: 10.1016/j.vaccine.2007.03.049. Epub 2007 Apr 20. PMID 17499406
- [Background] Smith JF, Brownlow M, Brown M, Kowalski R, Esser MT, Ruiz W, Barr E, Brown DR, Bryan JT. Antibodies from women immunized with Gardasil cross-neutralize HPV 45 pseudovirions. Hum Vaccin. 2007 Jul-Aug;3(4):109-15. doi: 10.4161/hv.3.4.4058. Epub 2007 Feb 24. PMID 17611417
- [Background] Ault KA; Future II Study Group. Effect of prophylactic human papillomavirus L1 virus-like-particle vaccine on risk of cervical intraepithelial neoplasia grade 2, grade 3, and adenocarcinoma in situ: a combined analysis of four randomised clinical trials. Lancet. 2007 Jun 2;369(9576):1861-1868. doi: 10.1016/S0140-6736(07)60852-6. PMID 17544766
- [Background] Giuliano AR, Lazcano-Ponce E, Villa L, Nolan T, Marchant C, Radley D, Golm G, McCarroll K, Yu J, Esser MT, Vuocolo SC, Barr E. Impact of baseline covariates on the immunogenicity of a quadrivalent (types 6, 11, 16, and 18) human papillomavirus virus-like-particle vaccine. J Infect Dis. 2007 Oct 15;196(8):1153-62. doi: 10.1086/521679. Epub 2007 Sep 17. PMID 17955433
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 1 received a 20/40/40/20 formulation of quadrivalent human papillomavirus (qHPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 2 received a 40/40/40/40 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 3 received a 80/80/40/80 formulation of quadrivalent human papillomavirus (qHPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the qHPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
- Placebo (mcg) (Aluminum Adjuvant) 225: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 4 received placebo containing 225 mcg of aluminum adjuvant per dose at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the qHPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
- Placebo (mcg) (Aluminum Adjuvant) 450: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 5 received placebo containing 450 mcg of aluminum adjuvant per dose at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the qHPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
- Extension 1: This group includes 241 international subjects, who either: (1) received placebo during the base study and continued in the Extension to receive a dose of GARDASIL (20/40/40/20 mcg formulation of qHPV vaccine) at Month 60 (plus 2 and 3 at Months 62 and 66, respectively, (2) received 3 doses of GARDASIL during the Base study and continued into the Extension to receive a fourth dose of GARDASIL at Month 60 for the purposes of investigating whether a fourth dose of vaccine (administered ~4.5 years following completion of a 3-dose primary regimen) induces HPV 6, 11, 16, and 18 antibody responses that characterize immune therapy.
- Extension 2: This group includes 17 subjects from the United States, who received placebo during the base study and received 3 doses of qHPV vaccine during the Extension, or received less than 3 doses of the qHPV Vaccine during the base study and completed the dose regimen during the Extension.
Period: Base Study (Day 1 to Month 7)
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450 | Extension 1 | Extension 2
Started | 290 | 284 | 292 | 146 | 146 | 0 | 0
Completed | 269 | 260 | 271 | 136 | 139 | 0 | 0
Not Completed | 21 | 24 | 21 | 10 | 7 | 0 | 0
Not completed — Randomized Not Vaccinated | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 6 | 6 | 4 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 3 | 2 | 3 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 9 | 12 | 4 | 3 | 0 | 0
Period: Long Term Follow-up (Month 7 toMonth 36)
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450 | Extension 1 | Extension 2
Started | 269 | 260 | 271 | 136 | 139 | 0 | 0
Completed | 137 | 245 | 251 | 57 | 57 | 0 | 0
Not Completed | 132 | 15 | 20 | 79 | 82 | 0 | 0
Not completed — Proceeded to Extension 1 | 114 | 0 | 0 | 69 | 75 | 0 | 0
Not completed — Lost to Follow-up | 6 | 8 | 5 | 4 | 3 | 0 | 0
Not completed — Moved | 3 | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 13 | 4 | 3 | 0 | 0
Period: Extension 1
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450 | Extension 1 | Extension 2
Started | 0 | 0 | 0 | 0 | 0 | 241 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 219 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 22 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 9 | 0
Not completed — Moved | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Extension 2
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450 | Extension 1 | Extension 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 17 (17 Participants continued into Extension 2 from Extension 1)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 1 received a 20/40/40/20 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
- Total: Total of all reporting groups
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450 | Total
Number analyzed (Participants) | 290 | 284 | 292 | 146 | 146 | 1158
Age, Continuous [Mean (Full Range); unit: years] | 20.2 [16 to 23] | 20.0 [15 to 24] | 20.1 [16 to 23] | 20.0 [16 to 23] | 20.1 [13 to 23] | 20.0 [13 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 290 | 284 | 292 | 146 | 146 | 1158
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 7 | 11 | 5 | 6 | 5 | 34
  Black | 25 | 32 | 27 | 12 | 7 | 103
  Hispanic American | 15 | 15 | 10 | 10 | 11 | 61
  Indian | 0 | 0 | 2 | 0 | 0 | 2
  Multi-racial | 13 | 9 | 6 | 7 | 4 | 39
  Native American | 2 | 4 | 2 | 0 | 1 | 9
  White | 228 | 213 | 240 | 111 | 118 | 910

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Injection Site Adverse Experiences
Time Frame: Days 1-5 following any vaccination visit
Population: All vaccinated subjects with adverse experience follow-up.
Measure: Number; unit: Participants
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450
Number analyzed (Participants) | 288 | 282 | 292 | 146 | 146
Participants | 247 | 248 | 266 | 107 | 115

2. Secondary Outcome: Incidence of HPV 6-, 11-, 16- or 18-related Persistent Infection or Disease (Cervical Intraepithelial Neoplasia, Vulvar Intraepithelial Neoplasia, Vaginal Intraepithelial Neoplasia, Adenocarcinoma in Situ, Cervical Cancer, and Genital Warts)
Time Frame: Through 36 Months
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative at Day 1 and PCR negative through Month 7 to the relevant HPV type, and must provide follow-up data after Month 7
Measure: Number; unit: Incidence per 100 person-years
Groups:
- Placebo (mcg) (Aluminum Adjuvant) 225 or 450 Combined: For the purposes of this outcome measure, the placebo groups (225 mcg and 450 mcg) were combined.
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Placebo (mcg) (Aluminum Adjuvant) 225 or 450 Combined
Number analyzed (Participants) | 235 | 233
Incidence per 100 person-years | 0.7 | 6.7
Statistical Analysis 1: Comparison: Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 vs Placebo (mcg) (Aluminum Adjuvant) 225 or 450 Combined; Test type: Superiority or Other; Vaccine Efficacy = 89.5, 95% CI [70.7 to 97.3] — Vaccine Efficacy (% relative risk reduction) Confidence Interval based on binomial tail probabilities and not from a dispersion parameter

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day 1 until Month 7. AEs were collected on the subject's vaccination report card daily for 14 days after each injection.
Description: Subjects were observed for 30 minutes after each vaccination. Temperatures were recorded for 5 days after each injection (4 hours after injection and daily for the next 4 days). At Months 2, 3, 6, and 7, subjects were solicited for any gynecological health concerns and any SAEs that had occurred.
Groups:
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 1 received a 20/40/40/20 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
  * There was one subject randomized to the quadrivalent HPV (Types 6, 11, 16, 18) L1 VLP vaccine 20/40/40/20 mcg group who received the 225 mcg aluminum adjuvant placebo at the third vaccination visit. This subject was not included in the counts reported in the Adverse Event tables. No SAEs were reported for this subject.
  * There was 1 patient that was randomized, but never vaccinated. As such, that patient is not included in this table.
- Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40: The Vaccination Period for the Base Study encompassed Day 1 through Month 7, during which time subjects in Group 2 received a 40/40/40/40 formulation of quadrivalent human papillomavirus (HPV) (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) vaccine at Day 1, Month 2, and Month 6.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the HPV 16 VLP Vaccine or placebo from completion of the Vaccination Period at Month 7 through Month 36.
  * There were 2 patients from the 40/40/40/40 group that were randomized, but were never vaccinated. As such, these 2 patients are not included in this table.
- Extensions: This group includes 241 international subjects, who either: (1) received placebo during the base study and continued in the Extension to receive a dose of GARDASIL (20/40/40/20 mcg formulation of qHPV vaccine) at Month 60 (plus 2 and 3 at Months 62 and 66, respectively, (2) received 3 doses of GARDASIL during the Base study and continued into the Extension to receive a fourth dose of GARDASIL at Month 60 for the purposes of investigating whether a fourth dose of vaccine (administered ~4.5 years following completion of a 3-dose primary regimen) induces HPV 6, 11, 16, and 18 antibody responses that characterize immune therapy.
  * Serious Adverse Events (SAEs) were collected during Extension 1 and Extension 2. Note that the N includes only the 241 subjects vaccinated during the Extension Periods; of the 258 subjects that entered either Extension, 17 subjects discontinued before being vaccinated and therefore are not included in this table.
Arm/Group | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 | Placebo (mcg) (Aluminum Adjuvant) 225 | Placebo (mcg) (Aluminum Adjuvant) 450 | Extensions
Serious Adverse Events (participants affected / at risk) | 3/288 | 0/282 | 2/292 | 0/146 | 3/146 | 1/241
Other Adverse Events (participants affected / at risk) | 245/288 | 247/282 | 263/292 | 105/146 | 114/146 | 180/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 (N=288) | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 (N=282) | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 (N=292) | Placebo (mcg) (Aluminum Adjuvant) 225 (N=146) | Placebo (mcg) (Aluminum Adjuvant) 450 (N=146) | Extensions (N=241)
Appendicitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Kidney infection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 20/40/40/20 (N=288) | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 40/40/40/40 (N=282) | Quadrivalent HPV (Types 6,11,16,18) L1 VLP Vaccine 80/80/40/80 (N=292) | Placebo (mcg) (Aluminum Adjuvant) 225 (N=146) | Placebo (mcg) (Aluminum Adjuvant) 450 (N=146) | Extensions (N=241)
Abdominal pain (Gastrointestinal disorders) | 13 | 14 | 16 | 5 | 9 | 0
Abdominal pain upper (Gastrointestinal disorders) | 10 | 16 | 8 | 7 | 3 | 0
Nausea (Gastrointestinal disorders) | 19 | 23 | 21 | 13 | 10 | 0
Fatigue (General disorders) | 26 | 8 | 23 | 9 | 9 | 0
Pyrexia (General disorders) | 30 | 37 | 41 | 13 | 16 | 14
Injection Site Erythema (General disorders) | 75 | 59 | 80 | 31 | 31 | 35
Injection Site Haematoma (General disorders) | 17 | 9 | 14 | 8 | 3 | 0
Injection Site Pain (General disorders) | 245 | 247 | 263 | 105 | 114 | 180
Injection Site Swelling (General disorders) | 80 | 74 | 95 | 23 | 29 | 46
Influenza (Infections and infestations) | 13 | 17 | 15 | 7 | 9 | 0
Nasopharyngitis (Infections and infestations) | 20 | 23 | 20 | 17 | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 10 | 8 | 9 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 6 | 4 | 7 | 9 | 0
Headache (Nervous system disorders) | 117 | 103 | 116 | 74 | 53 | 60
Dysmenorrhoea (Reproductive system and breast disorders) | 10 | 8 | 13 | 15 | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 10 | 17 | 11 | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.